CLINICAL TRIAL: NCT01012180
Title: Parents With Bipolar Disorder: Relationship of Adaptation to Own Illness With Risk Perception and Coping With Perceived Risk to a Child
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910007; 10-HG-N007
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-06-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Adaptation; Parents; Risk; Coping; Survey
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Bipolar disorder is a common mood disorder that affects 1% to 2% of the population. Individuals with bipolar disorder tend to have periods of mania that are characterized by extra energy, very poor judgment or unrealistic beliefs about their thoughts and abilities, and an inability to complete thoughts and tasks; as well as major depressive episodes. The range and frequency of symptoms in affected individuals can vary greatly. Most individuals have cyclical symptoms and spend more time in a normal mood state than in an overtly symptomatic state.
* Relatives of individuals with bipolar disorder have an increased risk for bipolar disorder and other mood disorders. Currently, risk assessment for recurrence of a mood disorder is based on family and medical histories; genetic testing has not proved particularly useful to date for assessing risks of a mood disorder.
* Despite its prevalence, there is limited research on coping with bipolar illness. No published studies have examined adaptation to living with bipolar disorder or risk for bipolar disorder. More specifically, though a positive family history is the most important known risk factor for bipolar disorder, there are no published studies about response to the threat of future illness onset in children, risk modification efforts undertaken by affected parents, or coping with the risk for illness in children.

Objectives:

* To examine parents appraisals of the impact and cause of bipolar disorder, and the association with their perceived risk for bipolar illness in their child and how they cope with their perception of risk to their child.
* To assess whether parents adaptation to their own illness is associated with coping with perceived risk to their child.
* To describe parents coping strategies related to perceived risk in their children.

Eligibility:

- Men and women at least 18 years of age who have been diagnosed with bipolar disorder and who have at least one biological child (30 years of age or younger). Participants must be a primary caregiver for their children.

Design:

* Participants in this study will take an online survey and answer questions about disease perceptions, coping strategies, and adapting to a diagnosis of bipolar disorder, addressing issues such as the following:
* Assessing the threat of bipolar disorder and coping with one s own illness.
* Optimism/pessimism of the individual coping with the illness.
* Perception of risk to a child, and coping with the perceived risk.
* Data from this study will not be shared with the participants/respondents.

DETAILED DESCRIPTION:
Though psychiatric disorders are extremely common and individuals with bipolar disorder have reproductive fitness approaching population rates, we know very little about the perceptions and coping of parents with bipolar disorder related to their at-risk children. Bipolar disorder is an etiologically-complex psychiatric disorder that is caused by a combination of genetic and environmental risk factors. This study proposes to assess perceptions of parents with bipolar disorder about their illness, response to illness threat, and concerns about their children s risks. We then propose to assess whether those appraisals are associated with the outcomes of coping strategies and adaption. As informed by the Transactional Theory of Stress and Coping, we propose to use a web-based survey to examine disease perceptions, coping strategies, and adaptation to the disorder. Respondents will be recruited through the National Alliance of the Mentally Ill (NAMI). The study is cross-sectional and the survey is composed of several valid and reliable scales to measure the constructs predicted to be involved in adaptation. Open-ended questions are included to help interpret results from the measures. Knowledge about parents perceptions and coping with their own illness and with risk to children may lead to studies of potential coping interventions. Ultimately, downstream studies may help to improve parents adaptation to their own condition and how successfully they are able to manage concerns about perceived risks to their child.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Have a diagnosis of bipolar disorder
* Be 18 years or older
* Be a biological parent of a child who is younger than 30 years old
* Be willing to participate in the survey
* The participant must be (or must have been) the primary caretaker for his or her child.

EXCLUSION CRITERIA:

* A participant must meet inclusion criteria.
* A participant s child cannot have been diagnosed with a mood disorder or other serious psychiatric disorder.
* A participant s child cannot have been adopted.
* The participant s child cannot be 30 years of age or older.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-10-23; Study Completion 2013-06-07

PRIMARY OUTCOMES:
Adaptation to bipolar disorder.

SECONDARY OUTCOMES:
Coping with perceived risk of bipolar to ones children.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland
  - NAMI Research Institute, Bethesda, Maryland

REFERENCES:
- [Background] Austin JC, Smith GN, Honer WG. The genomic era and perceptions of psychotic disorders: genetic risk estimation, associations with reproductive decisions and views about predictive testing. Am J Med Genet B Neuropsychiatr Genet. 2006 Dec 5;141B(8):926-8. doi: 10.1002/ajmg.b.30372. PMID 16958030
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744